CLINICAL TRIAL: NCT00190411
Title: Prevention of Vascular Complications by BetaBlocker Treatment in Vascular Ehlers-Danlos Syndrome
Brief Title: Celiprolol in Patients With Ehlers-Danlos Syndrome, Vascular Type
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: Aventis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: P010309
Record Dates: First submitted 2005-09-13; First posted 2005-09-19 (Estimated); Last update posted 2013-01-16 (Estimated); Status verified 2007-03

CONDITIONS: EHLERS-DANLOS SYNDROME, TYPE IV, AUTOSOMAL DOMINANT; CHROMOSOME 2q31.2 DELETION SYNDROME
Keywords: Arteries; ultrasonography; Ehlers Danlos syndrome; Cardiovascular disease; beta adrenergic antagonists
MeSH Terms: conditions — Ehlers-Danlos Syndrome, Type IV; Chromosome 2q31.2 Deletion Syndrome; Ehlers-Danlos Syndrome; Cardiovascular Diseases | interventions — Celiprolol

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment (Experimental): Celiprolol
  Interventions: Drug: celiprolol; Drug: Control

INTERVENTIONS:
Drug: celiprolol — celiprolol
  Other Names: celiprolol? Dose ranging 100 to 400 mg, dose adaptation; every 6 months by increment of 100 mg, based on tolerance
Drug: Control — Untreated controls excluding betablockers

SUMMARY:
Ehlers-Danlos syndrome vascular type (EDS-IV) is caused by a genetic defect of collagen type III. Patient die (median 40 yrs) of vascular complications. There is no treatment. We showed that arteries are thin and overloaded in this patients. We test the protective effect of celiprolol on cardiovascular events in a 5 years, randomized, PROBE design

DETAILED DESCRIPTION:
100 patients with verified EDS-IV syndrome are included. Patients are randomized to either celiprolol (50 to 400 mg BID)or no treatment. Patients who are not randomized enter a longitudinal survey of events. The hypothesis is a 50% reduction in the occurrence of cardiovascular events under treatment, assessed by a blinded, independent events committee.

ELIGIBILITY:
Inclusion Criteria:

* Proven disease,
* No betablocker at inclusion if previous CV event

Exclusion criteria:

Criteria of not inclusion for the RIGHTEOUS group:

* Patient having already presented an arterial break or a dissection and treated(handled) by bétâ-blocking(surrounding).
* Against indication in the use of CELIPROLOL:
* Unchecked cardiac insufficiency by the treatment
* cardiogenic shock
* BAV of 2nd and 3rd not sailed degrees
* angor of Prinzmetal
* disease of the sine
* bradycardia
* pheochromocytoma untreated
* low blood pressure
* sentimentality in the CELIPROLOL
* Antecedent of anaphylactic reaction
* myasthenia
* treatment by FLOCTAFENINE ( Idarac), Sultopride ( interactions ) In these two cases, the patient can be included in the group followed by troop.

Criteria of not inclusion for both groups:

* Refusal to participate in the study.
* Impossibility to move.
* Pregnancy
* Woman in age to procreate without means of effective contraception.

Ages: 15 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2003-10; Primary Completion 2011-04 (Actual); Study Completion 2011-04 (Actual)

PRIMARY OUTCOMES:
reduction in the rate of major cardiovascular events in the treated group during a 5 years follow-up | during de study
  reduction in the rate of major cardiovascular events in the treated group during a 5 years follow-up

SECONDARY OUTCOMES:
Tolerance, effect of drug on arterial parameters : diameter, IMT, stiffness. | during the study
  Tolerance, effect of drug on arterial parameters : diameter, IMT, stiffness.

CONTACTS AND LOCATIONS:
Overall Officials: Pierre BOUTOUYRIE, MD,PhD, Principal Investigator — Assistance Publique - Hôpitaux de Paris

REFERENCES:
- [Derived] Ong KT, Perdu J, De Backer J, Bozec E, Collignon P, Emmerich J, Fauret AL, Fiessinger JN, Germain DP, Georgesco G, Hulot JS, De Paepe A, Plauchu H, Jeunemaitre X, Laurent S, Boutouyrie P. Effect of celiprolol on prevention of cardiovascular events in vascular Ehlers-Danlos syndrome: a prospective randomised, open, blinded-endpoints trial. Lancet. 2010 Oct 30;376(9751):1476-84. doi: 10.1016/S0140-6736(10)60960-9. Epub 2010 Sep 7. PMID 20825986